CLINICAL TRIAL: NCT03997669
Title: The Diagnosis and Mechanism of Pleural Effusion
Status: Completed | Type: Observational
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Yang Jin, Professor, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Other Study IDs: 001
Record Dates: First submitted 2019-01-22; First posted 2019-06-25 (Actual); Last update posted 2021-11-16 (Actual); Status verified 2021-11

CONDITIONS: Pleural Diseases
MeSH Terms: conditions — Pleural Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The blood and pleural effusions if there is any, will be collected and detected
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- experimental group: patients with malignant pleural effusion
  Interventions: Other: Collection of pleural effusion
- control group: patients with benign pleural effusion
  Interventions: Other: Collection of pleural effusion

INTERVENTIONS:
Other: Collection of pleural effusion — Detection of pleural effusion

SUMMARY:
The diagnosis, treatment and mechanism of pleural diseases

DETAILED DESCRIPTION:
The diagnosis and treatment of benign and malignant pleural effusions, the mechanisms of pleural diseases

ELIGIBILITY:
Inclusion Criteria:

Patients with pleural effusion, who has not been treated

Exclusion Criteria:

Patients with pleural effusion, who has already been treated

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with pleural effusion
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
overall survival | 1 years
  the percentage of people in a group who are alive after a year for malignant pleural effusion

CONTACTS AND LOCATIONS:
Overall Officials: Jinshuo Fan, MD, Study Director — Key Laboratory of Respiratory Diseases of the Ministry of Health
Locations (1):
- Jinshuo Fan, Wuhan, State..., China

IPD SHARING:
Plan to Share IPD: Undecided